CLINICAL TRIAL: NCT00965211
Title: Evaluation of the HBDL Coil Transcranial Magnetic Stimulation (TMS) Device - Safety and Feasibility Study for the Treatment of Tourette Syndrome.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMS HBDL
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Tourette's Syndrome; Obsessive Compulsive Disorder
Keywords: Tourette's, OCD, dTMS, YGTSS, YBOCS, supplementary motor cortex; Tourette's syndrome and Obsessive compulsive disorder
MeSH Terms: conditions — Tourette Syndrome; Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: HBDL-coil Repetitive Deep Transcranial magnetic stimulation (rdTMS) — a session of rdTMS includes 4 cycles of 5 minutes of stimulation at a frequency of 1 Hz to the supplementary motor cortex and then a 2 minute recess.each subject would undergo 5 sessions a week for 4 weeks.

SUMMARY:
This is an open study.approximately 20 patients diagnosed with tourette's syndrome and under pharmAcological or psychotherapy treatments will participate.patients will be recruited from Schneider hospital and all his extensions. subjects would undergo rTMS (repetitive Transcranial Magnetic Stimulation) for five days a week, for four weeks,and will be clinically evaluated in order to monitor for improvement.

We anticipate a significant reduction in symptoms severity at the end of the treatment compared to study entry.

DETAILED DESCRIPTION:
Tourette's syndrome is a developmental neuropsychiatric disorder which is characterized by stereotypical motor and verbal bursts that are called Tics.

There is a small number of treatments that are available for the disorder, most of them are pharmacological agents that have serious side effects and are not very efficient in treating it.

In this current study we are attempting to find a better solution for the treatment of tourette syndrome using deep Transcranial magnetic stimulation(dTMS) technology.our region of interest for stimulation is the supplementary motor cortex (SMA). earlier superficial TMS studies focusing on the SMA have shown promising results. In theses studies clinical improvement was evident after two weeks of treatment, and for some of the subjects it was even maintained for a period of 3 months.we are using a similar protocol of TMS stimulation used in a study by Mantovani et al (2006).The protocol includes bilateral stimulation to the SMA at 110% of the motor threshold of the Abductor Policies Brevis and at a frequency of 1 Hz. each session is comprised of four cycles of 5 minutes of stimulation and a 2 minute recess.approximately 20 patients diagnosed with tourette syndrome and under pharmAcological or psychotherapy treatments will participate. patients will be recruited from Shnider hospital and all his extensions subjects would undergo rTMS sessions for five days a week, for four weeks, using the HBDL dTMS coil. this coil is capable of producing a magnetic field in deeper parts of the cerebral cortex, and for that reason we believe that it can produce better clinical outcomes then superficial TMS coils (such as the figure 8) used in past studies.

Clinical evaluation includes Yale-Brown Obsessive Compulsive Disorder Scale (YBOCS) , Yale Global Tic Severity rating Scale (YGTSS), Clinical Global Impression (CGI), Beck Depression Inventory (BDI), Symptoms Check List (SCL-90), Social Adaptation Self evaluation Scale (SASS), Hamilton Depression Rating Scale (HDRS-24), Hamilton Anxiety Rating Scale (HARS-14), Beck Depression Inventory (BDI) .These evaluation will be conducted on study entry, 2 weeks after study entry, at the end of the treatment phase and at a 2 week follow up visit (a total of four times). Further more, clinical evaluation will be administrated at Schneider hospital, while treatments are conducted at the cognitive lab at Shalvata hospital.

Our main objective is to observe a reduction in the severity of the symptoms post treatment in comparison to pre treatment, using the YGTSS as the main outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Men and woman between the ages of 18-55
* Diagnosed as suffering from tourette's syndrome according to the DSM IV, as determined by a senior psychiatrist on the basis of the Structured Clinical Interview for DSM-IV Axis I
* pharmocological treatment stays constant for the duration of the study
* Gave informed consent for participation in the study

Exclusion Criteria:

* Electroconvulsive therapy (ECT) less than 9 months prior to screening.
* Attempted suicide in the past year.
* History of seizure or heat convulsion.
* History of epilepsy or seizure in first degree relatives.
* History of head injury.
* History of any metal in the head (outside the mouth).
* Known history of any metallic particles in the eye, implanted cardiac pacemaker or any intracardiac lines, implanted neurostimulators, surgical clips or any medical pumps.
* History of frequent or severe headaches.
* History of migraine.
* History of hearing loss.
* Known history of cochlear implants
* Pregnancy or not using a reliable method of birth control.
* Inadequate communication with the patient.
* Under custodial care.
* Participation in current clinical study or clinical study within 30 days prior to this study.
* A significant physical illness which is not balanced.
* an addiction to psychoactive drugs in the last year or psychoactive substance abuse in the last month without addiction.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-09; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
The Yale Global Tic Severity rating Scale (YGTSS) | At study entry and every 2 weeks since then. total of 4 evaluation

SECONDARY OUTCOMES:
Yale-Brown Obsessive Compulsive Disorder Scale (YBOCS) | At study entry and every 2 weeks since. A total of 4 evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Eiran Vadim Harel, MD, Principal Investigator — Shalvata MHC
Locations (1):
- Shalvata Mental Health Center, Hod HaSharon, Israel